CLINICAL TRIAL: NCT00412516
Title: Long-Term Assessment at 24 Months Post-Vaccination of the Non-Inferiority of the Concurrent Administration of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine and Measles Vaccine to Measles Vaccine Given Alone
Brief Title: Determining Long-Term Safety and Efficacy of Japanese Encephalitis Vaccine When Given With Measles Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: JEV02
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Encephalitis, Japanese B
Keywords: Japanese Encephalitis; Japanese B Encephalitis; Japanese B Viral Encephalitis; Viral Encephalitis, Japanese B
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Other): JE live attenuated SA 14-14-2 vaccine then measles vaccine after one month
  Interventions: Biological: Live attenuated SA 14-14-2 vaccine
- Group 2 (Experimental): JE live attenuated SA 14-14-2 vaccine and measles vaccine concurrently
  Interventions: Biological: Live attenuated SA 14-14-2 vaccine
- Group 3 (Other): Measles vaccine then JE live attenuated SA 14-14-2 vaccine after one month
  Interventions: Biological: Live attenuated SA 14-14-2 vaccine

INTERVENTIONS:
Biological: Live attenuated SA 14-14-2 vaccine — Live attenuated SA 14-14-2 vaccine coadministered with live measles vaccine (experimental Group)

SUMMARY:
The previously conducted JEV01 study looked at the immunogenicity and safety of the concurrent administration of Japanese Live Attenuated SA 14-14-2 and measles vaccines at the one month post vaccination time point. The purpose of the JEV01 study was to help ensure the safety of SA 14-14-2 simultaneously administered with measles vaccine, paving the way for its use in routine EPI programs. As a follow-on to JEV01, this study will enroll those infants who received both vaccines and completed the JEV01 study. This study, however, will provide crucial data to help ensure the long-term immunogenicity of the concurrent administration of these vaccines and provide valuable information to determine the use of these vaccines in routine immunization programs. This study is planned because in the original protocol for JEV01, long-term data points were not included. The hypothesis is that children who receive JE live attenuated SA 14-14-2 vaccine and measles vaccine at the same time have long-term (24 and 36 months post vaccination) protection against these diseases at the same level as those who receive the vaccines at different intervals.

DETAILED DESCRIPTION:
Japanese encephalitis is the leading cause of viral neurological disease and disability in Asia. The severity of sequelae, together with the volume of cases, make JE the most important cause of viral encephalitis in the world. Approximately 3 billion people-including 700 million children-live in Asian areas at risk for JE. JE most commonly infects children between the ages of 1 and 15 years, and can also infect adults in areas where the virus is newly introduced. More than 50,000 cases are reported annually and cause an estimated 10,000 to 15,000 deaths. This figure is believed to represent only a small proportion of the disease burden that actually exists.

An effective vaccine has existed since 1941, but has not reached the poorest countries in Asia. During the 60 years that the vaccine has been available, JE has infected an estimated 10.5 million children, resulting in more than 3 million deaths and more than 4 million children living with long-term disabilities. Control of this disease has been limited due to poor disease surveillance, a limited and unstable vaccine supply, lack of guidance and programmatic support for immunization, and limited advocacy.

A successful vaccine should be safe, efficacious, affordable, administered in a single dose, and easily incorporated into the routine Expanded Programmes on Immunization (EPI) programs.

This trial is designed to determine the potential interference between the measles vaccine and the Japanese encephalitis vaccine at 12, 24, and 36 months post-vaccination. As these vaccines will be used in routine EPI systems at the same time, similar to how measles and yellow fever vaccine (also a Flavivirus) are administered, it is imperative to collect long-term data showing that neither vaccine interferes with seroconversion of the other when co-administered.This information will help to ensure subject safety and facilitate programmatic efficiency, reducing the number of immunization visits for both parents and health care workers.

ELIGIBILITY:
Inclusion Criteria:

* Participant was enrolled in the JEV01 study previously conducted at RITM.
* Participant completed his/her vaccination schedule for the JEV01 study previously conducted at RITM.
* Participant's blood test results from JEV01 study indicate that he/she had seroconverted to measles vaccination.
* Participant's parents or legal guardian are/is willing to provide signed informed consent.

Exclusion Criteria:

* Participant was withdrawn from the JEV01 study for any reason.
* Receipt of immune globulin or other blood products within 6 months of study (JEV02) entry or receipt of injected or oral corticosteroids or other immune modulator therapy (except routine vaccines) within 4 weeks of study (JEV02) entry.
* Any condition that in the opinion of the investigator, would interfere with the evaluation of the study objectives.

Ages: 20 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 519 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvacion Gatchalian, MD, Principal Investigator — Research Institute for Tropical Medicine (RITM)
Locations (1):
- Research Institute for Tropical Medicine (RITM), Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: SA 14-14-2 followed by measles vaccine one month later
- Group 2: Measles and SA 14-14-2 given concurrently
  Live attenuated SA 14-14-2 vaccine: Live attenuated SA 14-14-2 vaccine coadministered with live measles vaccine (experimental Group)
- Group 3: Measles vaccine followed by SA 14-14-2 one month later
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 93 | 212 | 214
Completed | 93 | 212 | 214
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all subjects enrolled in the study
Groups:
- Group 2: Measles and SA 14-14-2 given concurrently
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 93 | 212 | 214 | 519
Age, Continuous [Mean (Standard Deviation); unit: months] | 20.6 (.4) | 20.6 (.4) | 20.6 (.4) | 20.6 (.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 114 | 117 | 277
  Male | 47 | 98 | 97 | 242
Weight (kg) [Mean (Standard Deviation); unit: units on a scale] | 10.2 (1.3) | 10.2 (1.6) | 10.2 (1.4) | 10.2 (1.4)
Height (cm) [Mean (Standard Deviation); unit: cm] | 78.7 (3.1) | 77.8 (3.8) | 78.1 (3.5) | 78.0 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Measles Seropositivity at 24 and 36 Months
Description: Seropositivity defined as an anti-MV IgG concentration of 120 mIU/mL determined with the Siemens ELISA
Time Frame: 24, 36 months post vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants seropositive
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 93 | 212 | 213
percentage of participants seropositive
  24 months post vaccination | 98.92 [94.15 to 99.97] | 95.75 [92.09 to 98.04] | 94.37 [90.37 to 97.06]
  36 months post vaccination | 94.62 [87.90 to 98.23] | 91.39 [86.73 to 94.82] | 91.04 [86.36 to 94.52]

2. Secondary Outcome: Measles Seropositivity at 12 Months
Description: Seropositivity defined as an anti-MV IgG concentration of 120 mIU/mL determined with the Siemens ELISA
Time Frame: 12 months post vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects seropositive
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 89 | 205 | 211
percentage of subjects seropositive | 87.64 [78.96 to 93.67] | 87.32 [81.97 to 91.55] | 87.2 [81.93 to 91.40]

3. Secondary Outcome: Seropositive Rate for Japanese Encephalitis (JE) Antibody in Infants in the Philippines Who Received Measles Vaccine (MV) Before, With, or After SA 14-14-2 JE Vaccination by Month After JE Vaccination.
Description: "Seropositive" defined as a person with neutralizing antibody against JE virus at a titer ≥ 1:10 in a 50% plaque-reduction neutralizing assay (PRNT-50)
Time Frame: 12 months, 24 months, and 36 months post vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects seropositive
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 93 | 212 | 214
percentage of subjects seropositive
  12 months post-JE vaccination | 90.4 [81.9 to 95.8] | 83.5 [77.6 to 88.4] | 86.1 [80.6 to 90.6]
  24 months post-JE vaccination | 81.1 [71.5 to 88.6] | 83.8 [77.8 to 88.6] | 80.7 [74.6 to 85.9]
  36 months post-JE vaccination | 79.3 [69.3 to 87.2] | 82.7 [76.7 to 87.6] | 81.9 [75.8 to 87.0]

4. Secondary Outcome: Geometric Mean Neutralizing Antibody Titer to Japanese Encephalitis (JE) Virus in Infants in the Philippines Who Received Measles Vaccine (MV) Before, With, or After SA 14-14-2 JE Vaccination by Month After JE Vaccination.
Description: Neutralizing antibody titer determined using a 50% plaque-reduction neutralizing assay (PRNT-50) for JE virus
Time Frame: 12, 24, 36 months post-JE vaccination
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 93 | 212 | 214
GMT
  12 months post-JE vaccination | 108 [70 to 167] | 83 [61 to 108] | 77 [60 to 98]
  24 months post-JE vaccination | 67 [46 to 99] | 64 [50 to 80] | 70 [54 to 92]
  36 months post-JE vaccination | 51 [37 to 71] | 47 [38 to 58] | 58 [45 to 73]

ADVERSE EVENTS:
Time Frame: Three years post vaccination
Description: Since no investigational products were administered to subjects during the course of this study, subjects were not actively monitored to detect adverse events (AEs). However, passive surveillance was maintained to note reports of events meeting the definition of a serious AE (SAE).
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 4/93 | 14/212 | 13/214
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=93) | Group 2 (N=212) | Group 3 (N=214)
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 1
Ascariasis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 3 | 3
Cholera (Infections and infestations) | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 3
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Viral rash (Infections and infestations) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Developmental delay (General disorders) | 0 | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All results communication must be reviewed and approved by the sponsor. The sponsor has 60 days to review results communications and provide comments.